CLINICAL TRIAL: NCT06237283
Title: Effects of Early Postoperative Showering After Coronary Artery Bypass Grafting Using Bilateral Internal Thoracic Artery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sejong General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BSH 2023-09-005
Record Dates: First submitted 2024-01-23; First posted 2024-02-01 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Wounds and Injuries; Wound Infection
MeSH Terms: conditions — Wounds and Injuries; Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early shower (Experimental): Start shower after drain removal
  Interventions: Behavioral: Early shower
- Late shower (No Intervention): Start shower after wound stitches are removed

INTERVENTIONS:
Behavioral: Early shower — Start shower after drain removal
  Arms: Early shower

SUMMARY:
The study to evaluate effects of early postoperative showering after coronary artery bypass grafting using bilateral internal thoracic artery

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Patients who underwent coronary bypass grafting with bilateral internal thoracic artery through median sternotomy
* Patients whose all drains or pacing wires are removed

Exclusion Criteria:

* Concomitant operation
* Redo-surgery
* prolonged intensive care unit stay (more than 4 days) due to serious complications after surgery
* open wounds
* active infection
* prolonged drains

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Rate of deep sternal wound infection | until 1 months after discharge
Rate of superficial sternal wound infection | until 1 months after discharge
Rate of wound dehiscence | until 1 months after discharge

SECONDARY OUTCOMES:
Patient satisfaction | at 1st outpatient clinic visit
  questionnaire
Rate of mortality | until 1 months after discharge
Rate of stroke | until 1 months after discharge
Rate of respiratory complications | until 1 months after discharge
Rate of bleeding requiring reoperation | until 1 months after discharge
Rate of low cardiac output syndrome | until 1 months after discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Bucheon Sejong Hospital, Bucheon-si, Gyeonggi-do, South Korea